CLINICAL TRIAL: NCT01989039
Title: IR, Inflammatory and Cardiovascular Markers in PCOS Among Obese and Non-obese Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, Taipei Medical University WanFang Hospital, Taipei Medical University WanFang Hospital
Other Study IDs: Hsu2013-TMU-JIRB201307021
Record Dates: First submitted 2013-10-21; First posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Polycystic Ovary Syndrome,; Insulin Resistance,
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
FPCOS is associated with an adverse cardiometabolic profile, consisting of increased total or central adiposity, increased insulin resistance and abnormal glucose metabolism. Low-grade chronic inflammation predicts cardiovascular outcomes and is observed in women with PCOS. However, obesity is also associated with increased inflammatory markers. Obesity is per se associated with increased adipose expression and plasma levels of leptin, lower expression of adiponectin, and elevated inflammatory markers. To study the insulin resistance、inflammatory markers and cardiovascular risk in women with PCOS, body weight status should be considered. Investigator therefore conduct this retrospective study to evaluate the insulin resistance、inflammatory and cardiovascular markers between PCOS and non-PCOS among obese and non-obese women.

ELIGIBILITY:
Inclusion Criteria:

* Women had been fulfilled with whole anthropometric measurements, clinic and biochemical survey about insulin resistance, cardiovascular and inflammatory markers.

Exclusion Criteria:

* women who had been diagnosed with malignant tumor, Asherman's syndrome, Mullerian agenesis, ovarian failure, hyperprolactinemia, and chromosomal anomalies;
* women who had had menarche less than 1 years before evaluation or who were older than 49;
* women who received hormones or drugs for major medical diseases within three months.

Ages: 13 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women had been fulfilled with whole anthropometric measurements, clinic and biochemical survey about insulin resistance, cardiovascular and inflammatory markers.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-05 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Studying the insulin resistance, inflammatory and cardiovascular markers in polycystic ovary syndrome among obese and non-obese women. | A retrospective study in 800 Taiwanese women medical records reviewed from 2009 to 2012, up to 4 years in Wan Fang Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Ming I Hsu, MD, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- WanFang Medical Center at Taipei Medical University, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Shen SH, Shen SY, Liou TH, Hsu MI, Chang YC, Cheng CY, Hsu CS, Tzeng CR. Obesity and inflammatory biomarkers in women with polycystic ovary syndrome. Eur J Obstet Gynecol Reprod Biol. 2015 Sep;192:66-71. doi: 10.1016/j.ejogrb.2015.06.022. Epub 2015 Jul 2. PMID 26177495
- [Derived] Chen CI, Hsu MI, Lin SH, Chang YC, Hsu CS, Tzeng CR. Adiponectin and leptin in overweight/obese and lean women with polycystic ovary syndrome. Gynecol Endocrinol. 2015 Apr;31(4):264-8. doi: 10.3109/09513590.2014.984676. Epub 2014 Nov 25. PMID 25423261